CLINICAL TRIAL: NCT06397092
Title: Anesthetic Management for Transapical Beating-heart Septal Myectomy (TA-BSM) in Patients With Hypertrophic Obstructive Cardiomyopathy (HOCM)：A Retrospective Analysis
Brief Title: Anesthetic Management for TA-BSM in HOCM
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wenlong Yao (101480), Associate professor and deputy chief physician, Tongji Hospital
Other Study IDs: TongjiHospital-Anes QQ03
Record Dates: First submitted 2024-04-07; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Transapical Beating-heart Septal Myectomy; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TA-BSM: The hypertrophic cardiomyopathy patients received TA-BSM
  Interventions: Procedure: transapical beating-heart septal myectomy

INTERVENTIONS:
Procedure: transapical beating-heart septal myectomy — The patients with hypertrophic cardiomyopathy undergoing TA-BSM

SUMMARY:
To retrospectively analyze the preoperative, intraoperative and postoperative anesthesia management of patients with hypertrophic cardiomyopathy undergoing TA-BSM in the investigators' hospital, and to provide clinical basis for the development of reasonable and standardized perioperative anesthesia program for these patients.

DETAILED DESCRIPTION:
Hypertrophic obstructive cardiomyopathy is an inherited cardiomyopathy. Such patients have significantly reduced mobility and quality of life, and are prone to sudden death in severe cases. According to conservative estimates, there are about 2 to 5 million patients with hypertrophic heart disease in China, and about 15 to 20 million patients in the world, which seriously threatens human health. The traditional surgical treatment is partial ventricular septal myectomy through thoracotomy, which is traumatic and difficult, with poor efficacy and high operative mortality in hospitals with little experience.

In order to solve this problem, professor Wei's team invented and developed a beating-heart myectomy device, and established the first transapical beating-heart septal myectomy (TA-BSM) with the aid of this device through the apical minimally invasive incision under the guidance of esophageal ultrasound. With the help of echocardiography, the position of the rotator can be monitored in real time, and the angle and thickness of the rotator can be determined to ensure the safe removal of the hypertrophic ventricular septum, so as to solve the problem of left ventricular outflow tract obstruction.

The team firstly completed 47 clinical trials from April to September 2022, with a surgical success rate of 97.9%. At 3-month follow-up, the median maximum pressure gradient of left ventricular outflow tract decreased from perioperational 86 mmHg to postoperational 19 mmHg , and 45 participants (95.7%) had complete remission of mitral regurgitation. All patients showed significant improvement or even disappearance of symptoms, and exercise capacity and quality of life were significantly improved.

Since TA-BSM is a new surgical method, there is no unified standard for anesthesia management and lack of evidence-based evidence. Therefore, the aim of this study is to retrospectively analyze the preoperative, intraoperative and postoperative anesthetic management of participants with hypertrophic cardiomyopathy undergoing TA-BSM, so as to provide clinical basis for formulating reasonable and standardized perioperative anesthesia programs for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertrophic cardiomyopathy
* American Society of Anesthesiologists (ASA) physical status classification I-III
* Undergoing TA-BSM

Exclusion Criteria:

* Cardiopulmonary bypass was used to assist the surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The information of all patients with hypertrophic cardiomyopathy undergoing TA-BSM in our hospital from April 2022 to January 2023 was extracted and screened according to the inclusion criteria and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Perioperative information 1 | During surgery, when use isoproterenol to provocate
  Heart reat
Perioperative information 2 | During surgery, when use isoproterenol to provocate
  Systolic arterial blood pressure
Perioperative information 3 | During surgery, when use isoproterenol to provocate
  Diastolic arterial blood pressure
Perioperative information 4 | During surgery, when use isoproterenol to provocate
  Mean arterial blood pressure
Perioperative information 5 | Immediately after the surgery
  The type of tracheal tube
Perioperative information 6 | Immediately after the surgery
  The usage of anaesthetic drugs
Perioperative information 7 | Immediately after the surgery
  The usage of cardiovascular drugs
Perioperative information 8 | Immediately after the surgery
  Intraoperative infusion volume
Perioperative information 9 | Immediately after the surgery
  Blood transfusion volume
Perioperative information 10 | Immediately after the surgery
  Blood loss

SECONDARY OUTCOMES:
Postoperative information 1 | Postoperative in 30 days
  Extubation time,
Postoperative information 2 | Postoperative in 30 days
  Postoperative pain score: Pain score evaluation was performed after surgery ( 0-10 stands for the degree of the pain, 0 for painless and 10 for twinge).
Postoperative information 3 | Postoperative in 30 days
  The usagen of analgesic drug
Postoperative information 4 | Postoperative in 30 days
  Postoperative complications
Laboratory tests information 1 | 7 days before surgery and 3 days after surgery
  The changes of hemoglobin (Hb)
Laboratory tests information 2 | 7 days before surgery and 3 days after surgery
  the changes of creatinine (Cr)
Laboratory tests information 3 | 7 days before surgery and 3 days after surgery
  the changes of albumin (Alb)
Laboratory tests information 4 | 7 days before surgery and 3 days after surgery
  the changes of cardiac uhrasonography findings

CONTACTS AND LOCATIONS:
Overall Officials: Wenlong Yao, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong Science and Technology University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No